CLINICAL TRIAL: NCT04998890
Title: A Randomized Controlled Trial of Adventure-based Cognitive Behavioural Intervention for University Students in Hong Kong
Brief Title: Improving Mental Health of Chinese University Students in Hong Kong: Adventure-based Cognitive Behavioural Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Jiayan Pan, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HKBU 22603717
Record Dates: First submitted 2021-08-06; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Adventure-based Cognitive Behavioral Intervention

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adventure-based cognitive behavioral intervention (Experimental): An adventure-based cognitive behavioral intervention program A 13-session adventure-based cognitive behavioral intervention program, including 6 lectures, 5 workshops and adventure training (one adventure day camp (2 sessions) and adventure activities in the beginning of each workshop). One session per week, 3 hours for each session. A variety of cognitive behavioral skills were taught in lectures and these skills were practiced in two groups (with appropriately 20 students in each group) in workshop to help students to apply these skills to cope with their own daily life stress. Skill briefing, case demonstration and debriefing, group sharing and discussion, in-class exercise and homework were used in the intervention program.
  Interventions: Other: adventure-based cognitive behavioral intervention
- Control group (No Intervention): No intervention of the adventure-based cognitive behavioral program

INTERVENTIONS:
Other: adventure-based cognitive behavioral intervention — The adventure-based cognitive behavioral intervention is a combination of cognitive behavioral therapy and adventure training. The intervention program is delivered in a 39-hour general education course entailed "Improving Mental Health for University Success" in a public university in Hong Kong. The program includes 6 lectures, 5 workshops, 5 adventure games and an adventure day camp. Students are divided into two groups in workshop to practise CBT skills to deal with their own issues.
  Arms: Adventure-based cognitive behavioral intervention

SUMMARY:
This study delivered an adventure-based cognitive behavioral intervention program to a group of Hong Kong university students. The program effectiveness was evaluated by a randomized controlled trial in reducing psychological distress and improving mental health of these students. The 3-month maintenance effect was also tested.

DETAILED DESCRIPTION:
University students are vulnerable to mental health problems due to the various challenges they have to face in university life. However, few studies have been conducted to evaluate the effectiveness of university counseling programs in Hong Kong. This project aims at developing and systematically evaluating a culturally adapted and adventure-based cognitive behavioral intervention (aCBI) program to decrease psychological distress and improve various mental health outcomes for Chinese university students in Hong Kong. The aCBI program was delivered in a form of general education course in a university setting. Randomized controlled trial (RCT) design was adopted. The program was evaluated its effectiveness in reducing psychological distress, perceived stress, depressive and anxiety symptoms, negative thoughts and negative emotions and increasing positive thoughts and positive emotions.

ELIGIBILITY:
Inclusion Criteria:

* be of Chinese nationality
* be studying in undergraduate programs at Hong Kong Baptist University (HKBU), as the aCBI program will be provided in the form of a general education course at this university
* have GHQ-12 scores of 2-10 (0-0-1-1) (i.e., mild to moderate levels of psychological distress)
* be willing to complete the entire process of the project.

Exclusion Criteria:

* have GHQ-12 scores of 0-1 (i.e., a low level of psychological distress) or 11-12 (i.e., a high level of psychological distress)
* have one or more psychosis
* have experienced severe depression with suicidal attempts/ideation in the past 3 months, as diagnosed by a psychiatrist or a clinical psychologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
General Health Questionnaire-12 | baseline: before the intervention program starts
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 | post-test: 1 month upon completion of the intervention program
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress
General Health Questionnaire-12 | 3-month follow-up test: 3 months after completion of the intervention program
  12-item rating scale for psychological distress, scale score ranges from 0-12, with a higher score indicating a higher level of psychological distress

SECONDARY OUTCOMES:
Perceived Stress Scale | baseline: before the intervention program starts
  10-item rating scale for perceived stress, scale score ranges from 0-4, with a higher score indicating a higher level of perceived stress
Perceived Stress Scale | post-test: 1 month upon completion of the intervention program
  10-item rating scale for perceived stress, scale score ranges from 0-4, with a higher score indicating a higher level of perceived stress
Perceived Stress Scale | 3-month follow-up test: 3 months after completion of the intervention program
  10-item rating scale for perceived stress, scale score ranges from 0-4, with a higher score indicating a higher level of perceived stress
Beck Depression Inventory | baseline: before the intervention program starts
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptoms
Beck Depression Inventory | post-test: 1 month upon completion of the intervention program
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptoms
Beck Depression Inventory | 3-month follow-up test: 3 months after completion of the intervention program
  21-item rating scale for depressive symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of depressive symptoms
Beck Anxiety Inventory | baseline: before the intervention program starts
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Beck Anxiety Inventory | post-test: 1 month upon completion of the intervention program
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Beck Anxiety Inventory | 3-month follow-up test: 3 months after completion of the intervention program
  21-item rating scale for anxiety symptoms, scale score ranges from 0-63, with a higher score indicating a higher level of anxiety symptoms
Automatic Thoughts Questionnaire | baseline: before the intervention program starts
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought.
Automatic Thoughts Questionnaire | post-test: 1 month upon completion of the intervention program
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought.
Automatic Thoughts Questionnaire | 3-month follow-up test: 3 months after completion of the intervention program
  14-item rating scale for positive and negative automatic thoughts, score ranges from 1-5 for the positive thought subscale and negative thought subscale, with a higher score indicating a higher level of positive/negative thought.
Chinese Affect Scale | baseline: before the intervention program starts
  20-item rating scale for positive and negative emotions, score ranges from 1-6 for positive emotion subscale and negative emotion subscale, with a higher score indicating a higher level of positive/negative emotion
Chinese Affect Scale | post-test: 1 month upon completion of the intervention program
  20-item rating scale for positive and negative emotions, score ranges from 1-6 for positive emotion subscale and negative emotion subscale, with a higher score indicating a higher level of positive/negative emotion
Chinese Affect Scale | 3-month follow-up test: 3 months after completion of the intervention program
  20-item rating scale for positive and negative emotions, score ranges from 1-6 for positive emotion subscale and negative emotion subscale, with a higher score indicating a higher level of positive/negative emotion
Chinese Making Sense of Adversity Scale | baseline: before the intervention program starts
  12-item rating scale for measuring sense-making coping, score ranges from "1" = "totally disagree" to "6" = "totally agree", with a higher score indicating a higher level of sense-making coping.
Chinese Making Sense of Adversity Scale | post-test: 1 month upon completion of the intervention program
  12-item rating scale for measuring sense-making coping, score ranges from "1" = "totally disagree" to "6" = "totally agree", with a higher score indicating a higher level of sense-making coping.
Chinese Making Sense of Adversity Scale | 3-month follow-up test: 3 months after completion of the intervention program
  12-item rating scale for measuring sense-making coping, score ranges from "1" = "totally disagree" to "6" = "totally agree", with a higher score indicating a higher level of sense-making coping.
Connor-Davidson Resilience Scale | baseline: before the intervention program starts
  25-item rating scale for measuring resilience, score ranges from "1" = "not true at all" to "5" = "true all the time". All the Item scores are summed up as a total score, with a higher score indicating greater resilience.
Connor-Davidson Resilience Scale | post-test: 1 month upon completion of the intervention program
  25-item rating scale for measuring resilience, score ranges from "1" = "not true at all" to "5" = "true all the time". All the Item scores are summed up as a total score, with a higher score indicating greater resilience.
Connor-Davidson Resilience Scale | 3-month follow-up test: 3 months after completion of the intervention program
  25-item rating scale for measuring resilience, score ranges from "1" = "not true at all" to "5" = "true all the time". All the Item scores are summed up as a total score, with a higher score indicating greater resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayan Pan, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Jiayan Pan, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No